CLINICAL TRIAL: NCT06639373
Title: The Road to Recovery Initiative (R2RI): an Observational Study of a Novel Model of Substance Use Care in a Canadian Setting
Brief Title: The Road to Recovery Initiative (R2RI)
Acronym: R2RI
Status: Recruiting | Type: Observational
Sponsor: BC Centre on Substance Use (Other)
Responsible Party: Sponsor
Other Study IDs: BCCSU-R2RI
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Substance-Related Disorders
Keywords: addiction; substance use; alcohol; opioids; harm reduction
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive; Harm Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- R2R Service Access: Individuals with a substance use disorder who access or are admitted to an R2R service
  Interventions: Other: Specialized clinical service access

INTERVENTIONS:
Other: Specialized clinical service access — A new model of addiction care that will offer comprehensive and coordinated service delivery

SUMMARY:
Despite substance use causing significant harms and cost to our health care system, British Columbia's (BC) current addiction treatment system remains under-resourced and fragmented. To address this, Providence Health Care (PHC) is expanding clinical addiction services as part of the Road to Recovery Initiative (R2R). The proposed study aims to generate novel data to promote fully evidence-informed and coordinated substance use care in BC and beyond. This study will explore substance use treatment trajectories, identify challenges and areas for growth in addiction health services, characterize important features of patients accessing care, and improve our provincial capacity to promptly tailor approaches to care in response to the substance use crisis.

DETAILED DESCRIPTION:
Since the declaration of a public health emergencies in Canada in 2016 and the United States in 2017 in response to rising overdose deaths, more than 400,000 Americans and 38,000 Canadians have died from drug overdoses. Within Canada, British Columbia (BC) shoulders a substantial burden of that loss, exceeding 13,000 overdose deaths since 2016. BC's unpredictable and toxic drug supply combined with the province's siloed and fragmented addiction treatment system are key contributors. The burden of disease, however, is not restricted to criminalized substances. The prevalence of alcohol misuse across Canada is at an unprecedented high, between 2015 - 2016 over 77,000 hospitalizations were attributed to alcohol related harms, with the highest rates again being observed in BC. Further, the substance use crisis has had a disproportional impact on Indigenous peoples as a consequence of colonialism and systemic racism. Accordingly, the provincial government and representative health organizations have urgently called for the development and implementation of a coordinated system of culturally safe substance use care that spans a continuum, ranging from harm reduction services to abstinence-based programming.

To address care gaps, Providence Health Care (PHC)-a regional health authority in the province of BC - in collaboration with the provincial government's Ministry of Mental Health and Addictions (MMHA), Vancouver Coastal Health (VCH) (another regional health authority) - is spearheading the Road to Recovery (R2R) Initiative, a first-of-its-kind model of substance use care. BC's existing substance use treatment system is comprised of both publicly- and privately-funded service providers in bed-based and outpatient settings. Quality and standards vary substantially between service providers, and inter-organizational communication is extremely limited. The R2R model of care seeks to address this by: (1) improving access to care through the creation of approximately 100 new substance use treatment beds; and (2) offering comprehensive substance use management along the entire care continuum (i.e., harm reduction, withdrawal management, bed-based recovery and outpatient longitudinal follow-up). A focus of the R2R model is inclusivity and honouring what matters most to individual patients to foster a safe recovery environment. Thus, close collaborations with Providence Health Care's Indigenous Wellness and Reconciliation (IWR) team and the BC Centre on Substance Use Indigenous Initiatives team has supported the integration of Indigenous cultural safety into the R2R model including through workflows and daily programming thereby meeting patients where they are at when they want and are in need of substance use care.

The proposed study will constitute a cohort of patients accessing substance use treatment services parallel to the phased operationalization of R2R in the VCH region. In this mixed-methods prospective cohort design, patients receiving R2R services will be observed through primary data collection at baseline and 12-month follow up via (1) interviewer-administered surveys and (2) semi-structured qualitative interviews over a 5-year study period. Participants will be asked to provide consent for the use of personal identifiers (i.e., a unique and persistent identifier issued to all provincial residents to access healthcare) to support secondary data-collection through (1) 30-day prospective follow-up from time of R2R admission using electronic medical record chart review, and (2) linkage annually to provincial health and administrative databases over a five-year follow-up period. A purposive sample of cohort participants will also be invited to participate in baseline and 12-month follow-up qualitative interviews.

Employing a convergent parallel design, quantitative and qualitative data collection will occur in parallel, of which results are later compared and related to one another. This will be an iterative process, as findings from each convergent analysis will inform adaptations and additions to data collection processes across implementation phases of R2R. The data will be leveraged to promote evidence-informed and coordinated substance use care through the integration of population and administrative data From cohort participant questionnaires, the investigators will gain an understanding of substance use treatment trajectories, identify challenges and areas for growth in addiction health services, characterize important features of patients accessing care, and improve our provincial capacity to promptly tailor approaches to care in response to the substance use crisis. Engaging with Indigenous participants for each study outcome will be critical to understanding the impact of building Indigenous cultural safety into the R2R model on relevant outcomes, and is supported by the IWR. Lastly, this work will support surveillance of evolving substance use trends, identify fixed and modifiable risk factors impacting substance use trajectories, as well build local, regional, and provincial partnerships to promptly respond to health challenges associated with the dynamic landscape of the substance use crisis. Collaboration with IWR throughout this work ensures that the collection and use of Indigenous data respects and upholds the principles of Indigenous data governance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able to provide written informed consent
* A resident of British Columbia
* Willing to comply with study procedures
* An individual who has accessed one or more R2R services

Exclusion Criteria:

* Individuals who have an acute, severe mental health condition (e.g., psychosis) precluding the opportunity to provide full informed consent
* Individuals who have an acute, severe medical condition (e.g., intubation) precluding the opportunity to provide full informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have accessed or been admitted to any R2R service.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2028-10-05 (Estimated); Study Completion 2033-10-05 (Estimated)

PRIMARY OUTCOMES:
Substance use patterns following R2R access | 1 year
  Metrics include frequency of use in the 12-months following R2R access
Health care utilization patterns following R2R access | 1 year
  Metrics include the count of hospitalizations, readmissions, and emergency department visits.
Substance use treatment trajectories | 1 year
  Metrics include completion status of substance use treatment programs within 12 months after R2R access.
Health among study participants over time | 1 year
  Metrics include count of comorbidities in the 12 months following R2R access.

CONTACTS AND LOCATIONS:
Overall Officials: Seonaid Nolan, MD, FRCPC, Principal Investigator — BC Centre on Substance Use
Locations (1):
- St. Paul's Hospital - Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website — https://www.bccsu.ca/road-to-recovery-study/